CLINICAL TRIAL: NCT03413852
Title: Treatment of Cerebral Arteriovenous Malformations With SQUID Liquid Embolic Agent - The CHOICE Study A Non-interventional, Prospective, Single-arm, International, Multicenter Study
Brief Title: Treatment of Cerebral Arteriovenous Malformations With SQUID Liquid Embolic Agent (CHOICE)
Acronym: CHOICE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Embo-Flüssigkeiten A.G. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-201701-SQUID
Record Dates: First submitted 2018-01-23; First posted 2018-01-29 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Arteriovenous Malformation
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SQUID non-adhesive liquid embolic agent — AVM embolization using SQUID non-adhesive liquid embolic agent

SUMMARY:
The objective of this study is to further establish that SQUID, an alternative liquid embolic agent with specific properties, is a safe and effective alternative in bAVM endovascular treatment strategy available to date. Therefore, the performance of SQUID will be documented and its safety of use will be confirmed in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient planned for one or multiple embolization sessions using SQUID to achieve occlusion of a previously untreated bAVM.*

  *Patients with a direct fistula or saccular/flow-related aneurysm previously treated with NBCA and/or coils may be included.
* Patient in whom the use of SQUID had been decided for an embolization alone or in association to neurosurgery or radiotherapy.
* Patient ≥18 years old.
* Patient or authorized representative dully informed and having no objection to the clinical data collection and medical file access. An informed consent form must be signed and dated whenever required by local legislation

Exclusion Criteria:

* Patient with bAVM not eligible for endovascular treatment.
* Patient with bAVM previously treated by embolization with other devices (Liquid embolic agent, NBCA, particles, and coils).*

  *Patients with a direct fistula or saccular / flow-related aneurysm previously treated with NBCA and/or coils may be included.
* Patient with bAVM previously treated with surgery or radiotherapy.
* Patient intended to undergo surgery and embolization during the same procedure at first embolization
* Patient with multiple bAVM or bAVM associated with dural arteriovenous Fistula*.

  *Patients with a direct fistula or saccular / flow-related aneurysm previously treated with NBCA and/or coils may be included.
* Patient presenting contra-indication to the use of SQUID according to the Instructions For Use.
* Intention to treat with any non-adhesive embolic liquid other than SQUID, or planned treatment with another non-adhesive embolic liquid over the course of the endovascular treatment phase.
* Patient planned for a total endovascular treatment phase duration exceeding 2 years.
* Patient participating in another clinical study evaluating another medical device, another procedure or a medication.
* Any condition or any situation that would prohibit the patient from coming to the investigational center for the follow-up as recommended by the study protocol between 3 and 6 months, or prohibit carrying out the telephone mRS assessments at 1 month after each embolization session and at 12 months after the end of the endovascular treatment phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients planned for embolization using SQUID to achieve occlusion of a previously untreated bAVM.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Score (mRS) | 3 to 6 months after the last embolisation session
  mRS is a scale used to measure the degree of handicap or dependence in daily activities of people who have suffered a stroke or other causes of neurological handicap.
  The scale ranges from 0 to 6, running from perfect health, without symptoms, to death.
  0 - No symptoms
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Death.

CONTACTS AND LOCATIONS:
Locations (19):
- University Hospital Antwerp, Edegem, Belgium
- Odense University Hospital, Odense, Denmark
- France (11):
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - Hospices Civils de Lyon, Bron
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Central, Nancy
  - Hôpital Lariboisière, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital Maison Blanche, Reims
  - CHU Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU Toulouse, Toulouse
- Germany (5):
  - Zentralklinikum Augsburg, Augsburg
  - Klinikum der Ruhr-Universität Bochum, Knappschaftskrankenhaus, Bochum
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Grosshadern, Munich
- San Gerardo Monza, Monza, Italy

IPD SHARING:
Plan to Share IPD: No